CLINICAL TRIAL: NCT06981130
Title: Supporting Antibiotic Stewardship in Primary Care Via Point-of-care Testing (POCT) for Acute Respiratory Tract Infections: An Interventional Study
Brief Title: ASPIRE II. Supporting Antibiotic Stewardship in Primary Care Via POCT
Acronym: ASPIRE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Wales (Other)
Collaborators: Cwm Taf University Health Board (NHS) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 322984
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acute Respiratory Infection
Keywords: ARI; MxA; CRP; NICE; POC; Primary Care

STUDY DESIGN:
Intervention Model Description: This study follows a single-group assignment model in which all participants presenting to general practice with symptoms of acute respiratory infection (ARI) undergo testing with a Point-of-Care (PoC) diagnostic device. The device measures C-reactive protein (CRP) and Myxovirus resistance protein A (MxA) to help differentiate between viral and bacterial infections. The intervention is applied uniformly, and outcomes such as test performance, diagnostic accuracy, clinician decision-making, and antibiotic prescribing behaviour are monitored prospectively. No randomisation or control arm is included, as the primary objective is to evaluate real-world clinical utility and diagnostic performance in a standard care setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Suspected with Acute Respiratory Infection (Other): Self-referred patients presenting ARI symptoms that have met the study inclusion criteria and have been recruited to the study.
  Interventions: Device: FebriDx Point of Care Test

INTERVENTIONS:
Device: FebriDx Point of Care Test — Patients self-referring to their GP practice with symptoms of acute respiratory infection (ARI) will receive the FebriDx point-of-care test during their clinical consultation.

SUMMARY:
Acute Respiratory Infections (ARIs) are a major contributor to antibiotic resistance, largely due to the over prescription of antibiotics driven by the subjective nature of clinical assessment. The ASPIRE II study aims to evaluate whether a Point-of-Care (POC) diagnostic test, utilising C-reactive protein (CRP) and Myxovirus resistance protein A (MxA) biomarkers to differentiate between viral and bacterial infections can support clinical decision-making and serve as an effective antimicrobial stewardship tool.

DETAILED DESCRIPTION:
In the first ASPIRE study, in which the POC test was taken after the consultation, 20 participants produced results in the ratio 10:7:3 (negative, bacterial, viral) with a 75% agreement to the antibiotic prescription given by the physician following face-to-face consultation. The observational ASPIRE I Study identified the need for a rapid POC test and highlighted areas in which the test could have been used to prevent over-prescribing of antibiotics when ARI's are identified as viral. The FebriDx POC test was also useful in identifying instances where antibiotics were not prescribed, when a bacterial infection is presented, proving an effective decision-making tool for antibiotic stewardship.

Antibiotic stewardship is fast becoming an essential measure to improve antibiotic prescribing by clinicians. Antibiotic stewardship not only presents a cost-effective strategy for the NHS but addressed the issue of antimicrobial resistance (AMR) and protects patients from harm caused by unnecessary antibiotic use.

The economic costs of antibiotic resistance are largely unknown, but it is anticipated that with an increased number of cases, effects to the economy could be severe. Infections and infectious diseases cost England & Wales an estimated £30 billion a year, with many cases of acute respiratory infections (Chaplin, 2017). POC diagnostic tests in a clinical setting could give clinicians the ability to distinguish between microbial and viral infections, providing a more informed decision to antibiotic prescribing.

The purpose of this study is to build upon data generated by the ASPIRE study that determined by retrospective evaluation, that a POC immunoassay can accurately be used to guide clinician's prescription decision. The ASPIRE 2 study will use the POC assay as an interventional decision tool prior to the GP's consultation of a suspected acute respiratory infection (ARI).

Upon clinical assessment, the current clinical practice prescribes antibiotics based on symptoms reported by the patient and a subjective review by the GP. This results in antibiotics being prescribed from an informed decision made by the clinician, based only from patient symptoms. The use of a dual marker immunoassay could guide informed decisions based on qualitative data and degree of infection using POC testing in Primary Care.

The POC assay uses a dual marker immunoassay to differentiate between a viral and bacterial infection. C-reactive protein (CRP) is raised in the blood stream in response to inflammation. CRP can be elevated in viral infections, but generally the rise is to higher levels in bacterial infections, especially severe bacterial infections. Another blood protein, the MxA protein, is selectively increased in people with viral infections and therefore has the potential to greatly enhance the rapid distinction between viral and bacterial respiratory infections.

NICE guidance from 2014 recommends the use of CRP POC test in the diagnosis and appropriate management of lower respiratory tract infections in adults aged 18 and over (excluding people with COPD) after clinical assessment whether antibiotics should be prescribed. The study POC assay data could be used as an effective tool alongside NICE guidelines to prescribe antibiotics based on CRP concentration where an infection may be viral. Recent clinical studies suggest the POC test is highly effective, yielding over 80% sensitivity and over 90% specificity when identifying bacterial and viral infections in adults (NICE, 2020).

ELIGIBILITY:
Inclusion Criteria:

* Subject >18 years of age.
* having new onset symptoms suggestive of acute respiratory infection (ARI within 7 days of seeking care: runny nose, nasal congestion, sore throat, cough, hoarse voice, shortness of breath) with or without fever.

Exclusion Criteria:

* Unable to provide informed consent.
* Undergoing end of life care.
* Immunocompromised or taking chemotherapy, oral steroids, or interferon.
* Receiving a live vaccine in the last 14 days.
* Taking antibiotics or antivirals in the last 14 days.
* Patients that have symptoms lasting more than 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Concordance between FebriDx result and clinician decision | End of recruitment period.
  The level of agreement between the FebriDx classification (viral or bacterial) and the clinician's initial diagnostic impression and treatment decision, to prescribe antibiotics or not.

SECONDARY OUTCOMES:
Sensitivity and Specificity of FebriDx vs. Clinical Judgement | End of recruitment period .
  Sensitivity (true positive rate) and specificity (true negative rate) of FebriDx in identifying bacterial or viral infections, using clinical decision as reference.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Kier Hardie Practice 3, Merthyr Tydfil, Rhondda Cynon Taff
  - Oaktree Surgery, Bridgend
  - Meddygfa Glan Cynon Surgery, Mountain Ash

IPD SHARING:
Plan to Share IPD: No